CLINICAL TRIAL: NCT05275296
Title: Prospective, Multi-center, Open-label, Non-inferiority, Randomized, Cotrolled Registration Trial of the Intracranial Visualized Stent for the Wide-necked Intracranial Aneurysms
Brief Title: Registration Trial of the Intracranial Visualized Stent for the Wide-necked Intracranial Aneurysms
Acronym: PROMISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MicroPort NeuroTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mermaid-2021-01-A
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Brain Diseases; Aneurysm; Intracranial Aneurysm; Cardiovascular Diseases
MeSH Terms: conditions — Brain Diseases; Aneurysm; Intracranial Aneurysm; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Microport NeuroTech Intracranial Visualized Stent
  Interventions: Device: Intracranial stent for wide-necked aneurysms
- control group (Active Comparator): LVIS™ and LVIS™ Jr
  Interventions: Device: Intracranial stent for wide-necked aneurysms

INTERVENTIONS:
Device: Intracranial stent for wide-necked aneurysms — Intracranial stent for wide-necked aneurysms

SUMMARY:
A registration trial of the Intracranial Visualized stent in the treatment of wide-necked intracranial aneurysms

ELIGIBILITY:
Inclusion Criteria:

* At the time of signing the informed consent form(ICF), the applicant shall be male or non-pregnant female, aged 18 to 80 years;
* Target aneurysms was diagnosed as intracranial wide-necked saccular aneurysms(neck ≥4mm, or body-neck ratio <2) by DSA/CTA/MRA；
* The diameter of the parent vessel should be 2.0 to 4.5mm;
* The target aneurysm should be suitable for stent-assisted coiling surgery and could be treated through one operation;
* Subject or its legal representative should be able to understand the purpose of this study, also agree to comply with protocol and sign the informed consent form voluntarily.

Exclusion Criteria:

* Subject whose mRS score was greater or equal to 3 during the clinical evaluation before enrollment;
* Subject with recurrent aneurysm which was already embolized through stent-assisted coiling surgery;
* Subject with multiple aneurysms that cannot be treated by single stent;
* Subject with aneurysm ruptured within 30 days;
* Subject who is not suitable for anesthesia or endovascular surgery;
* Subject with significant stenosis of the parent arterty(>50%)
* Subject who underwent major sugical procedure (such as internal fixation for limb fractures, tumor resection, surgery for vital organs, etc.) within 30 days before signing the ICF or would underwent major sugical procedure 60 days after signing the ICF;
* Subject who is currently participating in a clinical trial of another drug or device which has not met the primary endpoint, or who are expexted to participate in a clinical trial of another durg or device;
* Subject with conditions or pathological changes which may interfere with the use of instrument, including but not limited to: carotid artery dissection, vasculitis, aortic dissection, etc;
* Subject who is contraindicated with stent-assisted coiling:

Subject with allergy to required anti-platelet and/or heparin medications required for treatment; Subject with allergy to radiographic contrast; Subject with allergy to Nitinol, platinum-tungsten, platinum-iridium alloy.

* Women who is pregnant or now breastfeeding;
* Subject with a life expectancy less than 12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Adequate occlusion rate of aneurysms | Time Frame: 360±60 days
  The Raymond-Roy intracranial aneurysm occlusion classification was used to assess the rate of aneurysm occlusion postoperatively or at the time of primary endpoint assessment (12 months). Occlusion rates were reported as Class I: complete occlusion; Class II: residual neck; Class III: residual aneurysm. Adequate occlusion rate includes Class I and Class II.

SECONDARY OUTCOMES:
Complete occlusion rate of aneurysms | Time Frame: 360±30 days
  The Raymond-Roy intracranial aneurysm occlusion classification was used to assess the rate of aneurysm occlusion postoperatively or at the time of primary endpoint assessment (12 months). Occlusion rates were reported as Class I: complete occlusion; Class II: residual neck; Class III: residual aneurysm. Complete occlusion rate includes Class I
Retreatment rate | Time Frame: 360±30 days
  Percentage of subjects who had aneurysm recurrence and underwent a secondary suergry during follow-up
Successful stent placement | Intraoperation
  Successful stent placement was defined as the stent was successfully released at the appropriate position, and covered the aneurysm's neck completely while the parent artery remained unobstructed postoperatively.
Incidence od in-stent stenosis (≥50%) | Time Frame: 360±30 days
Incidence of device-relared stroke or death | perioperative
Incidence of ipsilateral stroke of neurological death | Time Frame: 360±30 days
Incidence of device-related severe adverse event | Time Frame: 360±30 days
Incidence of aneurysm rupture | Time Frame: 360±30 days

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China